CLINICAL TRIAL: NCT03060733
Title: Helicobacter Pylori Sample Collection Protocol POST-THERAPY
Brief Title: Helicobacter Pylori Sample Collection Protocol Post Therapy Subjects
Status: Completed | Type: Observational
Sponsor: DiaSorin Inc. (Industry)
Collaborators: ICON Clinical Research (Industry)
Responsible Party: Sponsor
Other Study IDs: POST-TREAT Z001
Record Dates: First submitted 2017-02-15; First posted 2017-02-23 (Actual); Last update posted 2019-02-07 (Actual); Status verified 2019-02

CONDITIONS: Helicobacter Pylori Infection; Gastric Ulcer; Nausea; Abdominal Pain; Weight Loss; Stomach Ulcer; Loss of Appetite; Bloating
MeSH Terms: conditions — Stomach Ulcer; Nausea; Abdominal Pain; Weight Loss; Anorexia | interventions — Aftercare

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Human Stool
Oversight: FDA-regulated Drug: No

INTERVENTIONS:
Other: Post-Therapy — Gastric biopsy tested by composite reference method (CRM) (histology, urease, culture) and stool sample

SUMMARY:
The primary objective is to obtain stool samples from post-therapy subjects already undergoing evaluation for an H. pylori infection by upper esophagogastroduodenoscopy (EGD) and gastric biopsy.

DETAILED DESCRIPTION:
Stools will be collected and tested, at a later date, in a clinical performance study with an investigational H. pylori antigen assay. This study will be coordinated by the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 22 years, either gender
* Subject previously diagnosed with H. pylori infection
* Subject received and completed FDA approved treatment option
* Minimum of 4 weeks to one year has lapsed after completion of FDA approved treatment option
* Subject with a post therapy positive result from a FDA cleared UBT or FDA cleared Fecal Antigen Test
* Subject will undergo EGD and gastric biopsy as part of routine care to measure H. pylori post-therapy response
* Biopsy is obtained from antrum and/or corpus and is tested by CRM
* At least two of the three CRM tests are performed
* Subject whose EGD with biopsy occurred ≤ 7 days prior to stool collection
* Willing and able to sign the IRB approved Informed Consent form for this study project

Exclusion Criteria:

* Subject with current severe H. pylori infection
* Subject ingested compounds that may interfere with detecting of H. pylori, e.g. 4 weeks for antibiotics and 2 weeks for Bismuth preparations or proton pump inhibitors prior to collection
* Pregnant or lactating
* Inability or unwilling to perform required study procedures
* Subject is unable or unwilling to provide informed consent

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects are evaluated for H. pylori infectious status prior to eligibility. Evaluation includes use of a diagnostic H. pylori test, such as, an FDA cleared UBT or an FDA cleared Fecal Stool Antigen. Infectious status must be determined positive for H. pylori for subject eligibility.
  Eligible subjects are undergoing EGD with biopsy for H. pylori infectious status after completion of therapy
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2018-05-14 (Actual); Study Completion 2018-05-14 (Actual)

PRIMARY OUTCOMES:
Helicobacter pylori Stool Collection | Through Study Completion, an average of 1 year
  In vitro diagnostic (IVD) device performance

CONTACTS AND LOCATIONS:
Locations (5):
- United States (4):
  - One (1) Location in California, Mission Hills, California
  - One (1) Location in Great Neck, New York, Great Neck, New York
  - One (1) Location in Ohio, Mentor, Ohio
  - One (1) Location in Houston, Texas, Houston, Texas
- One (1) Location in Bologna, Italy, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided